CLINICAL TRIAL: NCT06335147
Title: PD1 Antibody Combined With mFOLFOX6 Neoadjuvant Therapy for Advanced Resectable Metastatic Colon Cancer，Single Arm, Multicenter Phase II Clinical Study
Brief Title: PD1 Antibody Combined With mFOLFOX6 Neoadjuvant Therapy for Advanced Resectable Metastatic Colon Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10IIT114
Record Dates: First submitted 2024-02-23; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serplulimab, mFOLFOX6 (Experimental): Serplulimab，200mg，iv，q2w，d1； mFOLFOX6（Oxaliplatin: 85 mg/m2，LV ：400mg/m2，Fluorouracil： 400mg/m2 d1，2400 mg/m2 continuous intravenous drip for 46-48 hours；q2w）
  Interventions: Drug: Serplulimab, mFOLFOX6

INTERVENTIONS:
Drug: Serplulimab, mFOLFOX6 — Serplulimab，200mg，iv，q2w，d1； mFOLFOX6（Oxaliplatin: 85 mg/m2，LV ：400mg/m2，Fluorouracil： 400mg/m2 d1，2400 mg/m2 continuous intravenous drip for 46-48 hours；q2w）
  Other Names: HLX10

SUMMARY:
Evaluate the efficacy and safety of PD1 monoclonal antibody combined with mFOLFOX6 neoadjuvant therapy for advanced resectable metastatic colon cancer with enriched pro-inflammatory pan macrophage subpopulations

DETAILED DESCRIPTION:
In this study, patients with advanced resectable metastatic colon cancer requiring neoadjuvant chemotherapy were selected, and colon cancer patients enriched with TNFSF10+CXCL10+ panTAMs subgroup were screened, and neoadjuvant chemotherapy was performed with PD-1 monoclonal antibody combined with chemotherapy. To evaluate the efficacy and safety of PD-1 monoclonal antibody combined with neoadjuvant chemotherapy in the treatment of special types of colon cancer.

All patients in this study were examined in the tumor microenvironment before treatment, and only patients enriched with TNFSF10+CXCL10+ panTAMs subgroup were enrolled in the study. Due to the long detection time, the patient received mFOLFOX6 chemotherapy for one week in the first cycle. If the test results meet the enriched proinflammatory panmacrophage subpopulation, patients can eventually be enrolled and receive PD-1 monoclonal antibody (Serplulimab, Srulimab) combined with mFOLFOX6 (oxaliplatin, fluorouracil) regimen, 2 weeks for 1 cycle. The primary radical resection was performed after 5 cycles of neoadjuvant therapy. Local treatment of liver/lung metastases was performed at the same time or at different times. Continue mFOLFOX6 chemotherapy for 4-6 cycles or CAPEOX regimen for 4 cycles within 1-2 months after surgery. Liver and lung metastases allow local treatment in any of these treatment cycles, including but not limited to radiofrequency ablation, particle implantation, radiation therapy, and surgery. At the end of postoperative adjuvant therapy, NED status was achieved. Then, regular follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Signed the inform consent
* Age >=18 years old, female and male
* Locally advanced or metastatic colorectal adenocarcinoma (including sig-ring cell carcinoma, mucinous adenocarcinoma, etc.) confirmed by pathology (histology or cytology)
* Enriched with proinflammatory panmacrophage subsets
* At least one measurable or evaluable lesion according to RECIST 1.1; Measurable lesions should not have received local treatment such as radiotherapy (Metastases can still be used as target lesions to evaluate efficacy after biopsy. Periintestinal lymph node imaging determines metastasis, allowing for a minimum diameter of ≥ 10mm, and can also be used as target lesions.)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* The life expectancy is ≥6 months；And according to the MDT in the hospital, only neoadjuvant chemotherapy is needed
* Hemoglobin content (HB) ≥ 90g/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L;Platelet count (PLT) ≥ 100 × 109/L (did not use interleukin-11 or TPO within 14 days);White blood cell count (WBC) ≥ 4.0 × 109/L (no use of granulocyte stimulating factor within 14 days).
* Total serum bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN); ALT and AST ≤ 2.5 × ULN;Cr ≤ 1.5 × ULN or creatinine clearance rate (CCr) ≥ 60ml/min, (Cockcroft Gault formula);Serum albumin ≥ 25 g/L (2.5 g/dL)
* For liver metastasis subjects, AST and ALT must be ≤ 5 x ULN, and white blood cells must be ≥ 4 × 109/L, platelets without blood transfusion ≥ 100 × 109/L, absolute neutrophil count (ANC) ≥ 1.5 without granulocyte stimulating factor treatment × 109/L, hemoglobin ≥ 90 g/L
* Doppler ultrasound evaluation: Left ventricular ejection fraction (LVEF) ≥ lower limit of normal value (50%).
* Adequate coagulation function, defined as international standardized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN;

Exclusion Criteria:

* Allergy to any investigational drug or its excipients, or a history of severe allergies, or contraindications to investigational drugs;
* Having a history of autoimmune diseases or being in an active phase;
* Symptomatic/Asymptomatic Brain Metastasis
* CT indicates clear ulcerative lesions or fecal occult blood positive for three or more consecutive times, and clinical considerations suggest the presence of gastrointestinal bleeding
* Abnormal thyroid function or taking thyroxine tablets
* Previously received allogeneic bone marrow transplantation or organ transplantation;
* Congenital pulmonary fibrosis, drug-induced pneumonia, organized pneumonia, or CT confirmed active pneumonia;
* HIV positive, active hepatitis B or C, active pulmonary tuberculosis;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response（pCR） | 1 month after resection
  pCR is defined as the percentage of participants in the analysis population who have a pathologic complete response

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1 month after resection
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by investigator.
2-year overall survival rate | 2-year
  Overall survival is defined as the time from randomization to death due to any cause
Incidence of Treatment-Emergent Adverse Events | up to 6 months
  All participants with treatment-related adverse events as assessed by National Cancer Institute Common Terminology Criteria for Adverse Event,Version 4.0(CTC AE4.0).

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, Principal Investigator — Henan Cancer Hospital

IPD SHARING:
Plan to Share IPD: No